CLINICAL TRIAL: NCT01324375
Title: Is Preoperative Pain Response Upon Tonic Heat Stimulation Predictive for Pain After Total Hip Arthroplasty?
Brief Title: Prediction of Pain in Total Hip Arthroplasty
Status: Completed | Type: Observational
Sponsor: Hvidovre University Hospital (Other)
Responsible Party: Principal Investigator, Troels Haxholdt Lunn, MD, Hvidovre University Hospital
Other Study IDs: H-2-2010-052, part 2
Record Dates: First submitted 2011-03-25; First posted 2011-03-29 (Estimated); Last update posted 2012-09-26 (Estimated); Status verified 2012-09

CONDITIONS: Pain, Postoperative
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood samples
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- THA (total hip arthroplasty): Patients undergoing THA, preoperatively heat tested
  Interventions: Device: heat pain test (Modular Sensory Analyzer, Somedic AB, Horby, Sweden).

INTERVENTIONS:
Device: heat pain test (Modular Sensory Analyzer, Somedic AB, Horby, Sweden). — pain during heat test preoperatively

SUMMARY:
In this consecutive, prospective cohort study the investigators evaluate if preoperative pain response upon heat stimulation is predictive for acute and subacute postoperative pain after total hip arthroplasty.

DETAILED DESCRIPTION:
The preoperative heat stimulation consists of short and long tonic heat stimulation. Pain response is evaluated with an electronic visual analog scale.

Furthermore the investigators evaluate other factors possibly predictable for acute and subacute postoperative pain after total hip arthroplasty - demographic factors, preoperative pain related factors, psychosocial factors (Hospital Anxiety and Depression Scale and Pain Catastrophizing Scale).

ELIGIBILITY:
Inclusion Criteria:

* Ethnic danes, above 18 years and able to give informed consent scheduled for primary, unilateral total hip arthroplasty

Exclusion Criteria:

* Bilateral/revision arthroplasty
* Disease affection central or peripheral nerve function
* Alcohol and medical abuse
* Daily use of opioids or glucocorticoids
* Malignancy
* BMI > 40
* Depression
* Dementia or other cognitive dysfunction

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergoing total hip arthroplasty (THA)
Sampling Method: Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2011-03; Primary Completion 2012-03 (Actual); Study Completion 2012-03 (Actual)

PRIMARY OUTCOMES:
Pain (from 0-24 hours after surgery) | 24 hours
  Pain assessed with the visual analog scale

SECONDARY OUTCOMES:
Pain (from day 1 to day 7 after surgery) | 7 days
  Pain assessed with the visual analog scale
Pain at day 14 after surgery | 14 days
  Pain assessed with the visual analog scale
Pain at day 30 after surgery | 30 days
  Pain assessed with the visual analog scale

CONTACTS AND LOCATIONS:
Overall Officials: Troels H Lunn, MD, Principal Investigator — Dep. of Anesthesiology, Hvidovre University Hospital
Locations (1):
- Dep. of Anesthesiology, Hvidovre University Hospital, Copenhagen, Hvidovre, Denmark